CLINICAL TRIAL: NCT07090993
Title: Behavior Development Training for Sustainable Nutrition for Nutrition and Dietetics Department Students: A Randomized Controlled Study
Brief Title: Behavior Development Training for Sustainable Nutrition
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betul Uner (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Betul Uner, Lecturer, MSc, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocol No: 240034
Record Dates: First submitted 2025-06-23; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Sustainable Nutrition; Sustainable Healthy Diet; Sustainable Food Consumption; Sustainable Lifestyles; Mediterranean Diet
Keywords: Mediterranean diet; RCT; sustainability; sustainable nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sustainable nutrition education (Experimental): sustainable nutrition education
  Interventions: Behavioral: sustainable nutrition education
- waiting list (No Intervention): No intervention is made during the study. At the end of the study, the same training given to the intervention group is applied to this group.

INTERVENTIONS:
Behavioral: sustainable nutrition education — The educational intervention applied to the experimental group was carried out in 12 sessions. The knowledge-attitude-behavior education model was adopted in the education sessions. The education program, which was created by obtaining expert opinions, consists of five basic topics and was carried out with the interactive education method.
  Sessions;
  1. Environmental effects during the production of animal and plant foods
  2. Production and environmental effects of processed foods
  3. Foods with low environmental impact and nutrition models
  4. What are food losses and wastes?
  5. Workshops
  6. Processing and storage of foods
  7. Consumption of local, regional and seasonal fruits, vegetables and fish
  8. The importance of sustainable nutrition and alternative protein sources
  9. Mediterranean diet model
  10. Preparing a shopping list
  11. Reading labels and nutritional content
  12. Watching a documentary on the harms of packaged foods on living beings and the environment
  Arms: sustainable nutrition education

SUMMARY:
The European Federation of Dietetic Associations (EFAD) recommends sustainable nutrition to create healthy societies. Sustainable nutrition models include the Mediterranean diet, vegetarian and vegan diets, the double pyramid model, and the Scandinavian diet.

The dilemma of food loss, waste, and hunger is one of the significant paradoxical problems faced in today's world. Food waste and wastage can become an environmental and economic problem if not managed properly.

It is stated that the difficulties in accessing animal protein will increase daily due to the increasing and continuing global population and negative environmental impacts.

A literature review revealed the lack of a randomized controlled trial on behavioral education for sustainable nutrition among university students. This study aims to educate Nutrition and Dietetics students about sustainable nutrition, food waste, and waste, to translate the information provided to students into behavioral behavior, and to contribute to the literature in this field. In this randomized controlled experimental study, the "Sustainable Nutritional Behavior Development Scale" and the "Mediterranean Diet Adherence Scale" will be administered face-to-face to healthy students actively studying in the Department of Nutrition and Dietetics at Muğla Sıtkı Koçman University's Faculty of Health Sciences, and their scores will be calculated.

Following the initial data collection process, students assigned to the experimental group will receive a 12-week training program based on the knowledge-attitude-behavior model (Bettinghaus, 1986). Students will be included in the Sustainable Nutritional Behavior Development Training Program, while the control group will not receive any intervention. After data collection, in accordance with ethical principles, students in the control group will receive the same training as students in the experimental group.

The collected study data will be analyzed using SPSS 20.0 statistical analysis software. The Kolmogorov-Smirnov test will be used to assess data normality. Findings regarding the students' individual characteristics will be analyzed using percentages, means, and standard deviations. The relationship between the independent variables of the control and experimental groups and the anthropometric measurement results and scale scores will be examined with appropriate statistical analyses.

DETAILED DESCRIPTION:
The term sustainable development was first used in the World Economic Development Commission (WCED) Brundtland 1987 report. The concept of sustainable development is based on three moral obligations: meeting human needs, ensuring social equality and respecting environmental limits (United Nations Turkey).

The ability of the atmosphere to transmit and retain heat is called the greenhouse gas effect. Agricultural production is among the reasons for the increase in greenhouse gases (Turkish Statistical Institute (TUIK), Greenhouse Gas Emission Statistics). The rapid increase in the world population has also caused the food sector to grow. The greenhouse gas formation caused by agricultural practices can be examined under three headings, grouped as animal husbandry, rice fields and other activities. Due to the increasing food demand, environmental pollution caused by animal production facilities has increased significantly as a result of the development of meat and dairy cattle, dairy industry and poultry farming.

Another factor affecting the greenhouse gas formation is the carbon and water footprint. A 3-fold increase in the carbon footprint level has been observed in Turkey in a 15-year period. Turkey is among the countries that may experience a drought problem (State Hydraulic Works (DSİ)). It is a fact that animal-based products require more water than plant-based products. This shows that the water footprint of animal-based nutrition models is higher than plant-based nutrition models. When the water footprint values of foods are examined, they are listed from the highest to the lowest as follows; beef, lamb, animal milk, nuts, butter, goat meat, cheese, legumes, eggs, oilseeds, cereals, fruits, and vegetables. It is predicted that there will be a water shortage due to increasing population and usage after 2030 (World Wildlife Fund (WWF)).

It is known that the preference of diet models that are known to have lower environmental impacts can play a key role in the concept of sustainability. The Food and Agriculture Organization (FAO) has put forward the concept of sustainable diet to emphasize the importance of the subject; It is defined as diets that have lower environmental impacts, are reliable in terms of nutrition and nutrition, and can ensure the continuity of a healthy life for future generations. The Livewell for Low Impact Food in Europe (LIFE) project, carried out by the World Wildlife Fund (WWF), which supports sustainable nutrition, consists of 6 basic rules. These rules are; increasing the consumption of vegetables and fruits, ensuring nutritional diversity, preventing food waste, reducing meat consumption, purchasing certified food, and reducing the consumption of foods high in fat, salt and sugar and sugary drinks.

The European Federation of Dietetic Associations (EFAD) recommends following sustainable diets in creating healthy societies. When the basic characteristics of a sustainable diet are examined, it is seen that vegetables and fruits with lower environmental impacts are predominant, and animal-based foods known to have higher environmental impacts are restricted. Sustainable nutrition models include the Mediterranean diet, vegetarian and vegan diet, double pyramid nutrition model and Nordic diet.

Mediterranean diet; It has been proven that it has significant effects on the environment in addition to its positive effects on human health, which has been used since the 1960s. It was understood in the 1990s that the ecological footprint of the foods consumed in the Mediterranean diet was much lower compared to the foods in Western-style diets. For this reason, the Mediterranean diet is considered a suitable diet type for sustainable nutrition.

Vegetarianism is defined as the frequent consumption of plant-based foods instead of animal-based foods. The diet in which red meat, chicken and fish are not consumed or are limited, and eggs, milk and dairy products are consumed optionally is called "vegetarianism". Veganism, one of the types of vegetarianism, is defined as a lifestyle that refuses to use animal-based food, cosmetics, clothing and all other by-products for some reasons. Recent studies have shown that plant-based nutrition has positive results in human health and that western-style diet models negatively affect planetary health, so it is among the sustainable nutrition models.

The double pyramid model is a sustainable nutrition model that supports the consumption of environmentally friendly and local foods created by the Barilla Food and Nutrition Center (BCFN) in Italy. This model states the inverse relationship between the foods consumed and the environmental impacts of those foods.

The traditional diet of Northern European countries is the Nordic Diet (ND) and is based on seasonal foods. While giving importance to taste, health and sustainability issues with ND, it is in harmony with regional food culture and eating habits. ND is recommended as an alternative to the Mediterranean diet. Excessive meat consumption has negative effects on both individual health and environmental health. The Nordic diet includes fruits and vegetables with low environmental impacts, wild herbs and game, fish and seafood, potatoes and cereals.

Food loss and waste and hunger dilemma is one of the important paradoxical problems experienced in the world today. While all losses occurring due to reasons such as problems in planning and food processing, operational, financial and technological problems throughout the food supply chain stages are defined as food losses; food waste is also defined as not consuming food due to reasons such as color, shape, excessive purchase, large portioning or throwing away at the consumer stage. It has been stated that the period when the highest amount of losses occur in Turkey is the agricultural production stage, which is one of the food supply chain stages, with a rate of 11.9%. In our country, it has been shown by the TÜİK report that fish and seafood are the least wasted and fruits and vegetables are the most wasted. A systematic review that supports the TÜİK report has indicated that fruits and vegetables are the most wasted nutrients in the National School Lunch Program. According to the results of a study evaluating household food waste, the reasons for waste include purchasing too much food, lack of shopping and cooking plans, and lack of knowledge in preserving and storing food. Food waste and waste can be an environmental and economic problem if not managed properly. Ways to combat food waste and waste can be listed as regular storage, anaerobic digestion, composting and creating animal feed.

It is stated that the difficulties in accessing animal-based protein will increase day by day due to the increasing and continuing world population and negative environmental effects. Environmental pollution, climate crisis, the decrease in agricultural activities due to increased migration to cities, the decrease in world resources and the increase in food waste reveal that sustainability should be included in nutrition.

When the literature was reviewed, no randomized controlled study was found on university students regarding behavioral training for sustainable nutrition. This study aims to educate students of the Nutrition and Dietetics department, who will be the future community nutrition experts, on sustainable nutrition and food waste and waste, to help students develop correct behaviors through educational activities provided, and to contribute to the literature in this field.

ELIGIBILITY:
Inclusion Criteria:

* To be a 2nd year student in the Department of Nutrition and Dietetics
* To be between the ages of 18-35
* To have no health problems

Exclusion Criteria:

* Being an active student
* Being a 1st, 3rd or 4th year student
* Having a diet that complies with sustainable nutrition models
* Having attended any training, conference, symposium on sustainable nutrition and/or received information on this subject in any way

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
The effect of sustainable nutrition education on adherence to the Mediterranean diet | The training takes an average of 12 weeks to complete.
  Participants' adherence to the Mediterranean diet will be assessed using the Mediterranean Diet Adherence Scale (MEDAS). Scale scores range from 0 to 14. A higher score indicates greater adherence to sustainable nutrition principles.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University/Muğla Training and Research Hospital Neurology Polyclinic, Muğla, Mentese, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR